CLINICAL TRIAL: NCT05473884
Title: CIVILIAN Study in Femoropopliteal Artery Occlusion Disease
Brief Title: Lesion Preparation in Femoropopliteal Artery Occlusion Disease
Acronym: CIVILIAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Xuanwu Hospital, Beijing (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Second Affiliated Hospital of Soochow University (Other); Qingdao Hiser Medical Group (Other)
Responsible Party: Principal Investigator, Bo Yu, MD, Professor, Shanghai Pudong Hospital
Other Study IDs: Shanghai-CIVILIAN
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Femoropopliteal Artery Occlusion; Atherosclerosis Obliterans; Lesion; Vascular; In-stent Restenosis
Keywords: femoropopliteal Artery Occlusion; debulking; drug-coated balloon; bail-out stenting; endovascular therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lesion preparation with POBA in femoropopliteal Artery occlusion: Patients with femoropopliteal artery occlusion were treated by plain old balloon angioplasty followed with DCB.
  Interventions: Device: conventional balloon
- lesion preparation with debulking devices in femoropopliteal Artery occlusion: Patients with femoropopliteal artery occlusion were treated by other lesion preparation devices, like Chocolate balloon, Shockwave balloon, TurboHawk, Jetstream and Rotarex and then followed by DCB.
  Interventions: Device: lesion preparation devices

INTERVENTIONS:
Device: lesion preparation devices — successful recanalization of femoropopliteal artery occlusion and then followed by lesion preparation devices and plain old balloon angioplasty
  Other Names: Chocolate balloon; Shockwave balloon; Rotarex; TurboHawk; Jetstream
  Groups: lesion preparation with debulking devices in femoropopliteal Artery occlusion
Device: conventional balloon — Lumen gain is achieved by plain old balloon angioplasty under working inflation pressure.
  Groups: lesion preparation with POBA in femoropopliteal Artery occlusion

SUMMARY:
Peripheral arterial disease (PAD) carries a significant global health burden, and can limit functional capacity and quality of life. Percutaneous transluminal angioplasty (PTA) for PAD is often associated with suboptimal outcomes due to complications following balloon inflation related to vessel trauma and flow limiting dissections that may require bailout stenting. Different strategies and techniques to enhance both acute and longer-term outcomes with drug-coated balloons (DCB) are needed. This is a national, prospective, multi-center, non-randomized, real-world study to evaluate the safety and efficacy of multiple vessel preparation strategies combined with drug-coating balloon (DCB) in Femoropopliteal Artery (F-PA) lesions.

DETAILED DESCRIPTION:
Femoropopliteal artery occlusive disease is a common type of peripheral arterial disease (PAD). Hitherto, endovascular treatment has been testified and advocated as the first-line treatment of femoropopliteal occlusive disease. However, the in-stent restenosis has been a major limitation of well long-term patency rate in this segment due to physiological and geometrical issues. The concept "leave nothing behind" is proposed, and some vessel preparation methods and devices, such as directional atherectomy, rotational atherectomy, laser atherectomy are developed. This is a national, prospective, multi-center, non-randomized study to evaluate the safety and efficacy of multiple vessel preparation strategies combined with drug-coating balloon (DCB) in Femoropopliteal Artery (F-PA) lesions. A total of 1000 patients will be included in approximately 8 sites. The study is designed to demonstrate the inferiority of different vessel preparation strategies in various fields under long-term follow-up.

ELIGIBILITY:
General Inclusion Criteria:

* Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed an Ethical Committee approved consent form
* Patient has a score from 2 to 5 following Rutherford classification
* Unilateral or bilateral F-P occlusive lesions (enrollment of one or both target limbs depend on operators)
* Complete recanalization followed by POBA, Chocolate PTA, Scoring PTA, Shockwave PTA, SilverHawk, TurboHawk, Jetstream, Angiojet, Laser and Rotarex

Angiographic Inclusion Criteria:

* TASC II-Type A/B/C/D
* Iliac inflow interventions can be done at the discretion of the investigator with standard balloon Percutaneous Transluminal Angioplasty (PTA)-less than 50% residual stenosis
* There is angiographic evidence of at least one-vessel-runoff (>10cm) to the foot

General Exclusion Criteria:

* Projected for major amputation of target limb (above ankle joint)
* Change to thrombectomy or bypass during operation
* Patients for whom antiplatelet therapy, anticoagulants, medium contrast, or thrombolytic drugs are contraindicated
* Patient has bleeding diathesis, coagulopathy, known hypercoagulable condition or refuses blood transfusion
* female patient with childbearing potential not taking adequate contraceptives or currently breastfeeding.
* Life expectancy of less than twelve months.
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.
* Patient presenting one of the following comorbid conditions: hemodialysis, elevated creatine levels (> 2.5mg/dl), recent MI or ischemic stroke occurrence (both within 30 days).
* Patient unwilling or unlikely to comply with Follow-Up schedule

Angiographic Exclusion Criteria:

* Testified for acute F-P arterial embolization
* Thromboangiitis obliterans
* Failed for recanalization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages Eligible for Study: 18 Years to 85 Years (Adult, Older Adult) Sexes Eligible for Study: All Accepts Healthy Volunteers: No
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from TLR | within 12 months post-procedure
  Percentage of participants with a 1-year TLR free survival
Incidence of complications | immediately following procedure (day 30)
  Procedure-related complications at day 30, defined as: procedure-related distal embolization, acute post-procedural target vessel thrombosis, bleeding, perforation, acute renal failure
Major adverse event | within 12 months post-procedure
  Major adverse events (MAE) rate at 1 year, defined as: Myocardial Infarction (MI), major amputation, all-cause mortality

SECONDARY OUTCOMES:
Technical Success | within 24 hours post-procedure
  Technical success, defined as the ability to cross the target lesion with the device, set up antegrade blood flow and leave residual stenosis <30%
Incidence of dissection and types | immediately following vessel preparation
  Dissection patterns according to the National Heart, Lung and Blood Institute classification system for the coronary artery. (Type A-F) (A) Type A has minor radiolucent areas, (B) type B is a linear dissection, (C) type C has contrast outside the lumen, (D) type D is a spiral dissection, (E) type E has persistent filling defects, and (F) type F is a total occlusion without distal antegrade flow
Incidence of Bailout stenting | immediately following vessel preparation and DCB angioplasty
  Bailout stenting, defined as stent implantation after vessel preparation and DCB including bare metal stents (BMS), covered stents and drug-eluting stents (DES)
Amputation Free Survival | within 12 months post-procedure
  Percentage of participants with a 1-year amputation free survival
Numbers of patients with Primary patency | within 3, 6, 12 months post-procedure
  Primary patency rate at 6, 12, 24 months as determined by Duplex ultrasound at six months, defined as a target vessel with <50% diameter stenosis (systolic velocity ratio no greater than 2.4), without occurrence of target lesion revascularization between the index procedure and follow-up control
Improvement of ABI | within 3, 6, 12 months post-procedure
  Increase of Ankle-Brachial Index (ABI) at 12, 24 months, defined as: an increase in ABI compared to baseline
Improvement of related symptoms | within 3, 6, 12 months post-procedure
  related symptoms could be identified as Rutherford classification from level 1-6.
  improvement in Rutherford classification compared to the pre-procedure Rutherford classification

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No